CLINICAL TRIAL: NCT02864511
Title: Nefertiti Lift for Neck Rejuvenation: Assessing Efficiency and Re-defining Patient Selection
Brief Title: Botulinum Toxin for Neck Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, samer jabbour, M.D., St Joseph University, Beirut, Lebanon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USJ-01
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Botulinum Toxin, Rejuvenation, Neck, Therapy

ARMS (1):
- Intervention group (Experimental)
  Interventions: Procedure: Nefertiti lift

INTERVENTIONS:
Procedure: Nefertiti lift
  Other Names: neck rejuvenation

SUMMARY:
The purpose of this study is to describe a safe and consistent technique for neck rejuvenation using botulinum toxin. This study will also evaluate the efficiency of the intervention and determine the patients that would benefit most.

DETAILED DESCRIPTION:
The abobotulinumtoxinA will be used for the Nefertiti lift The abobotulinumtoxinA will be prepared by adding 2.5 cc of normal saline to a 500-unit Dysport© (Ipsen Ltd, Berks, UK) vial Preinjection frontal, oblique and lateral patient pictures will be taken (at rest and with contraction)

Injection points:

* A series of 4 injection points 1-2 cm apart on a horizontal line under the mandible posterior to the hypothetical line were the nasolabial fold meets the mandible
* If present, injection of each platysmal band every 2 cm with 2 to 4 injection points per band (Injection of platysmal band will be done by holding the band between 2 fingers and injecting intramuscularly) For all injection points 5 units per point of abobotulinumtoxinA will be used

A maximum of 125 units of abobotulinumtoxinA will be allowed for the global neck treatment

Follow up will be done at 15 days for retouching or for post op pictures if no retouching is needed. if retouching is needed post injection pictures will be taken 10 days post retouching

Retouching: each residual platysmal band will be reinjected every 2 cm with 2 to 4 injection points per band (Injection of platysmal band will be done by holding the band between 2 fingers and injecting intramuscularly) (5 units per point of abobotulinumtoxinA will be used)

A total of 30 patients will be recruited

ELIGIBILITY:
Inclusion Criteria:

Female patients presenting to our clinic for neck rejuvenation who:

* Were deemed nonsurgical candidates for neck rejuvenation
* Were not willing to undergo invasive surgical procedures
* Had a medical contraindication to surgery

Exclusion Criteria:

* Patients with lower face botulinum toxin injection in the past 12 months
* Patients with resorbable lower face fillers injection in the past 12 months
* Patients with previous permanent lower face fillers injection
* Pregnant patients
* Lactating patients
* Patients with preexisting neuromuscular conditions (myasthenia gravis, Eaton Lambert syndrome)
* Patients using medication that could potentiate the effect of botulinum (ex: aminoglycoside antibiotics)
* Patients with sensitivity to botulinum toxin or human albumin

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Neck volume using a validated scale from the Summit Scale II (1) | 15-25 days post treatment
  The assessment will be done by 2 plastic surgeons and 1 dermatologist. Pre and post injection scores will be calculated by the independent evaluators based on the photographic scale . The 3 evaluators will be blinded to the pre or post injection status of the photos
  No Sagging
  Mild Sagging
  Moderate Sagging
  Severe Sagging
  Very Severe Sagging
Jowls at rest using a validated scale from the Summit Scale II (2) | 15-25 days post treatment
  The assessment will be done by 2 plastic surgeons and 1 dermatologist. Pre and post injection scores will be calculated by the independent evaluators based on the photographic scale . The 3 evaluators will be blinded to the pre or post injection status of the photos
  No Sagging
  Mild Sagging
  Moderate Sagging
  Severe Sagging
  Very Severe Sagging
Marionette lines at rest using a validated scale from the Summit Scale II (3) | 15-25 days post treatment
  The assessment will be done by 2 plastic surgeons and 1 dermatologist. Pre and post injection scores will be calculated by the independent evaluators based on the photographic scale . The 3 evaluators will be blinded to the pre or post injection status of the photos
  No visible folds: continuous skin lines
  Shallow but visible folds with slight indentation
  Moderately deep folds, clear feature at normal appearance, but not when stretched
  Very long and deep folds, prominent facial feature
  Extremely long and deep folds; detrimental facial appearance
Oral commissures at rest using a validated scale from the Summit Scale II (2) | 15-25 days post treatment
  The assessment will be done by 2 plastic surgeons and 1 dermatologist. Pre and post injection scores will be calculated by the independent evaluators based on the photographic scale . The 3 evaluators will be blinded to the pre or post injection status of the photos
  No Downturn
  Mild Downturn
  Moderate Downturn
  Severe Downturn
  Very Severe Downturn
Platysmal bands at maximal contraction using a validated scale (4) | 15-25 days post treatment
  The assessment will be done by 2 plastic surgeons and 1 dermatologist. Pre and post injection scores will be calculated by the independent evaluators based on the photographic scale . The 3 evaluators will be blinded to the pre or post injection status of the photos
  No relevant prominence of platysmal bands
  Mild prominence of platysmal bands
  Moderate prominence of platysmal bands
  Severe prominence of platysmal bands
  Very severe prominence of platysmal bands
Platysmal bands at rest using a validated scale (5) | 15-25 days post treatment
  The assessment will be done by 2 plastic surgeons and 1 dermatologist. Pre and post injection scores will be calculated by the independent evaluators based on the photographic scale . The 3 evaluators will be blinded to the pre or post injection status of the photos
  No platsymal bands visible at rest
  Mild platysmal bands evident at rest. Bands do not appear along the full length of the neck.
  Mild platysmal bands evident along the full length of the neck at rest, less than 5 mm of elevation from the surrounding tissue.
  Moderate platsymal bandsvisible at rest along the full length of the neck, elevation at least 5 mm from the surrounding tissue.
  Severe platsymal bands along the full length of the neck at rest, elevation at least 5 mm from the surrounding tissue, with additional soft tissue ptotic banding present laterally
Mandibular definition change with maximal contraction will be assessed by a 2-point scale | 15-25 days post treatment
  The assessment of the pre-injection photos will be done by 2 plastic surgeons and 1 dermatologist
  Mandibular contour does not worsen with platysmal contraction
  Mandibular contour worsen with platysmal contraction

SECONDARY OUTCOMES:
Investigators Global Aesthetic Improvement Scale | 15-25 days post treatment
  Improvement in Overall appearance (global neck, jowls, skin laxity, platysmal bands, mandibular contour), as assessed by the investigators using the Global Aesthetic Improvement Scale (GAIS). GAIS will be completed based on photographic assessment comparing post-treatment photos taken at day 15-25 post intervention to baseline photos, to assess overall aesthetic improvement. The GAIS is a 5-point scale (1-5) as follows:
  1. Very Much Improved: optimal cosmetic results
  2. Much Improved: marked improvement in appearance from initial condition but not completely optimal
  3. Improved: obvious improvement in appearance from initial condition but additional treatments are advised
  4. No Change: the appearance is the same as the original condition
  5. Worse: the appearance is worse from the original condition
Subject Global Aesthetic Improvement Scale | 15-25 days post treatment
  Improvement in Overall appearance (global neck, jowls, skin laxity, platysmal bands, mandibular contour), as assessed by the subject using the Global Aesthetic Improvement Scale (GAIS). GAIS will be completed based on a live assessment of the subject with a mirror in hand for real time assessment and and a photographic assessment comparing post-treatment photos taken at day 15-25 post intervention to baseline photos, to assess overall aesthetic improvement. The GAIS is a 5-point scale (1-5) as follows:
  1. Very Much Improved: optimal cosmetic results
  2. Much Improved: marked improvement in appearance from initial condition but not completely optimal
  3. Improved: obvious improvement in appearance from initial condition but additional treatments are advised
  4. No Change: the appearance is the same as the original condition
  5. Worse: the appearance is worse from the original condition
Patient satisfaction | 15-25 days post treatment
  Patient satisfaction will be determined by a questionnaire completed at 15-25 days post-treatment. Subjects will indicate how satisfied they are on a 4-point scale (1-4) as follow:
  1. Very Satisfied
  2. Satisfied
  3. Dissatisfied
  4. Very Dissatisfied.
Patient willingness to repeat the procedure | 15-25 days post treatment
  Patient willingness to repeat the procedure will be assessed by a simple question with a Yes or No response
Patient willingness to recommend the procedure | 15-25 days post treatment
  Patient willingness to recommend the procedure to a friend will be assessed by a simple question with a Yes or No response
Assessment of Pain during treatment | At the day of the procedure
  Subjects' pain during the treatment will be recorded using a validated Numeric Rating Scale (0-10), with 0 representing no pain and 10 representing the worst pain possible

CONTACTS AND LOCATIONS:
Locations (1):
- Hotel Dieu De France, Beirut, Aschrafieh, Lebanon

REFERENCES:
- [Background] Sattler G, Carruthers A, Carruthers J, Flynn TC, Geister TL, Gortelmeyer R, Hardas B, Himmrich S, Jones D, Kerscher M, Mohrmann C, Narins RS, Pooth R, Rzany B, Buchner L, Benter U, Breitscheidel L, de Maio M. Validated assessment scale for neck volume. Dermatol Surg. 2012 Feb;38(2 Spec No.):343-50. doi: 10.1111/j.1524-4725.2011.02253.x. PMID 22316190
- [Background] Narins RS, Carruthers J, Flynn TC, Geister TL, Gortelmeyer R, Hardas B, Himmrich S, Jones D, Kerscher M, de Maio M, Mohrmann C, Pooth R, Rzany B, Sattler G, Buchner L, Benter U, Breitscheidel L, Carruthers A. Validated assessment scales for the lower face. Dermatol Surg. 2012 Feb;38(2 Spec No.):333-42. doi: 10.1111/j.1524-4725.2011.02247.x. PMID 22316189
- [Background] Carruthers A, Carruthers J, Hardas B, Kaur M, Goertelmeyer R, Jones D, Rzany B, Cohen J, Kerscher M, Flynn TC, Maas C, Sattler G, Gebauer A, Pooth R, McClure K, Simone-Korbel U, Buchner L. A validated grading scale for marionette lines. Dermatol Surg. 2008 Nov;34 Suppl 2:S167-72. doi: 10.1111/j.1524-4725.2008.34366.x. PMID 19021675
- [Background] Geister TL, Blessmann-Gurk B, Rzany B, Harrington L, Gortelmeyer R, Pooth R. Validated assessment scale for platysmal bands. Dermatol Surg. 2013 Aug;39(8):1217-25. doi: 10.1111/dsu.12240. Epub 2013 May 7. PMID 23650974
- [Background] Gupta S, Biskup N, Mattison G, Leis A. Development and Validation of a Clinical Assessment Tool for Platysmal Banding in Cervicomental Aesthetics of the Female Neck. Aesthet Surg J. 2015 Aug;35(6):NP141-6. doi: 10.1093/asj/sju160. PMID 26229133